CLINICAL TRIAL: NCT04312555
Title: Efficacy of Alprostadil as an Adjuvant Therapy With Indirect Angiosomal Revascularization in Patients With Critical Limb Ischemia.
Brief Title: Alprostadil as an Adjuvant Therapy With Indirect Angiosomal Revascularization in Critical Limb Ischemia.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seif Eleslam Abdelhafiz Tawfik Ali, Resident doctor at Vascular & Endovascular surgery department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alprostadil with CLI
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Critical Limb Ischemia
Keywords: CLI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Alprostadil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Alprostadil — Alprostadil intravenous administration. (0.5 mg/1ml of Alprostadil + 49cm saline 0.9%) and 4 cm direct intravenously / 8 hours

SUMMARY:
The aim of this study is to assess the efficacy of Alprostadil (Prostaglandin E2) as adjuvant therapy after failure of direct but indirect angiosomal revascularization in patients with critical limb ischemia.

DETAILED DESCRIPTION:
In large number of elderly patients aged between 50 and 75 years, the arterial disease is prevalent (1%-7%). It has a significant impact on the quality of life. Pain, fear of limb loss, increased inactivity, and poor lifestyle choices which finally ended by disability. Disability in turn makes communities and counties carry more efforts and charges.

The incidence of critical limb ischemia (CLI) is increasing, and diabetic patients are especially prone to developing ischemic and neuro-ischemic foot ulcers. Twelve to 25% of diabetic patients may develop a foot lesion over time. Diabetic patients often present with more extensive tissue loss compared to non-diabetic patients. The importance of revascularization of the lower limb in patients with CLI has been well established, and expedited revascularization is mandatory once an ischemic foot ulcer is detected.

Although there is still a role for surgical bypass, over the last several decades the use of endovascular techniques has become more frequent. This development has been made possible by the evolution of endovascular devices and operator skills. The less-invasive endovascular approach is the preferred treatment method, especially in the frail diabetic patient with multiple comorbidities. Incisional wound healing in diabetic patients can also be problematic. In both open and endovascular revascularization there is a clear difference of approach in patients with CLI caused by inflow disease (iliac, femoral, and popliteal disease) and those with (additional) infrapopliteal involvement. Whereas in above-the-knee disease, it is clear that flow in the stenotic or occluded segment needs to be re-established, in below-the-knee (BTK) disease, potentially three vessels can be revascularized, and this poses a therapeutic dilemma. Choosing the correct target for revascularization can present a critical, complex issue in challenging cases, especially when multilevel arterial disease is present. Revascularization can be accomplished by using two approaches: "complete" revascularization (one vessel is better than none, two to three vessels are better than one) or "wound-related" revascularization. With CLI, the healing of an ulcer is blood-flow-dependent and the goal of treatment should be to get the best possible blood supply to the foot (direct revascularization). In practice this is not always feasible, and in order to guide the choice of which BTK vessel should be revascularized, the angiosome concept has been proposed, based on the idea that specific anatomical regions are perfused by specific arteriovenous bundles.

Prostaglandins are potent vasoactive agents with wide variety of other actions - vasodilatation, fibrinolysis and inhibition of platelet aggregation. PG infusion therapy may show a promising results in patients where such new reconstructive procedures are not feasible or failed and also as an adjunctive when there is a residual ischemia after the revascularization procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 40 years.
* Subject with chronic limb ischemia [Rutherford classification 4, 5 & 6].
* Subject failed to direct revascularization.
* Subject is able and willing to comply with the protocol and to adhere to the follow-up requirements.
* Subject has provided written informed consent.

Exclusion Criteria:

* Subject's age less than 40.
* Imminent or foreseeable amputation
* Subject already had a major amputation on the affected extremity
* Subject has emergent ischemic lesion [such as gas forming infection].
* Subject has a known hypersensitivity or contraindication to anticoagulants, anti-platelets, or contrast media, which is not amenable to pre-treatment.
* Subject has a known hypersensitivity or contraindication to Alprostadil.
* Subject is not in the position to be primarily revascularized or refuses surgery.
* Acute ischemia and peripheral vascular disorders of inflammatory or immunologic origin
* Neuropathic or venous ulcers
* Already using vasoactive medication or prostaglandins
* Treatment with prostanoids within 3 months prior to inclusion

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Patency | 3 months
  Maintaining vessel patency without restenosis or need for re-intervention
Major Adverse Limb Events (MALE) | 3 months
  repeated endovascular therapy, surgical revision, or major amputation during follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Elnaggar, Dr, Principal Investigator — Assiut University; Hassan Bakr El-Badawy, Prof, Study Chair — Assiut University; Mohamed Elsagheer Elhewwy, Prof, Study Director — Al-Azhar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kroger K, Hwang I, Rudofsky G. Recanalization of chronic peripheral arterial occlusions by alternating intra-arterial rt-PA and PGE1. Vasa. 1998 Feb;27(1):20-3. PMID 9540428
- [Background] Bucci M, Iacobitti P, Laurora G, Cesarone MR. [Analysis of costs and results of prostaglandin (PGE1 alpha-cyclodestrin) therapy of peripheral arterial diseases]. Minerva Cardioangiol. 1998 Oct;46(10 Suppl 1):9-15. Italian. PMID 10658439
- [Background] Palena LM, Garcia LF, Brigato C, Sultato E, Candeo A, Baccaglini T, Manzi M. Angiosomes: how do they affect my treatment? Tech Vasc Interv Radiol. 2014 Sep;17(3):155-69. doi: 10.1053/j.tvir.2014.08.004. PMID 25241316
- [Background] Neville RF, Sidawy AN. Surgical bypass: when is it best and do angiosomes play a role? Semin Vasc Surg. 2012 Jun;25(2):102-7. doi: 10.1053/j.semvascsurg.2012.04.001. PMID 22817860
- [Background] Iida O, Soga Y, Hirano K, Kawasaki D, Suzuki K, Miyashita Y, Terashi H, Uematsu M. Long-term results of direct and indirect endovascular revascularization based on the angiosome concept in patients with critical limb ischemia presenting with isolated below-the-knee lesions. J Vasc Surg. 2012 Feb;55(2):363-370.e5. doi: 10.1016/j.jvs.2011.08.014. Epub 2011 Nov 1. PMID 22051875
- [Background] Soderstrom M, Alback A, Biancari F, Lappalainen K, Lepantalo M, Venermo M. Angiosome-targeted infrapopliteal endovascular revascularization for treatment of diabetic foot ulcers. J Vasc Surg. 2013 Feb;57(2):427-35. doi: 10.1016/j.jvs.2012.07.057. Epub 2012 Dec 7. PMID 23219512
- [Background] Alexandrescu V, Hubermont G. Primary infragenicular angioplasty for diabetic neuroischemic foot ulcers following the angiosome distribution: a new paradigm for the vascular interventionist? Diabetes Metab Syndr Obes. 2011;4:327-36. doi: 10.2147/DMSO.S23471. Epub 2011 Aug 22. PMID 21969804